CLINICAL TRIAL: NCT03261141
Title: Correlation Between The Arabic Pediatric Voice Related Quality of Life (PV-RQOL), The Auditory Perceptual Assessment and Acoustic Analysis of Voice in Dysphonic Children
Brief Title: Correlation Between (PV-RQOL), The Auditory Perceptual Assessment and Acoustic Analysis of Voice in Dysphonic Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Fathy, principal investigator, Assiut University
Other Study IDs: PV-RQOL in Dysphonic children
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-08

CONDITIONS: Dysphonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group sixty three children: 1. severity and character of dysphonia APA using a modified GRBAS scale which gives scores as regard the degree and severity of dysphonia and its character.
  2. Acoustic Analysis of voice : which is Computerized Speech Laboratory analysis of voice that gives the following measures jitter (%), shimmer (dB), and harmonic to noise ratio (H/N).
  3. the degree of social ,emotional ,functional and physical disturbance ,if present in those children with voice disorders by application of The Arabic Pediatric Voice Related Quality of Life (PV-RQOL).
  Interventions: Combination Product: (PV-RQOL),(APA) ,Acoustic analysis
- control group sixty three children: 1. severity and character of dysphonia (APA using a modified GRBAS scale which gives scores as regard the degree and severity of dysphonia and its character.
  2. Acoustic Analysis of voice : which is Computerized Speech Laboratory analysis of voice that gives the following measures jitter (%), shimmer (dB), and harmonic to noise ratio (H/N).
  3. the degree of social ,emotional ,functional and physical disturbance ,if present in those children with voice disorders by application of The Arabic Pediatric Voice Related Quality of Life (PV-RQOL).
  Interventions: Combination Product: (PV-RQOL),(APA) ,Acoustic analysis

INTERVENTIONS:
Combination Product: (PV-RQOL),(APA) ,Acoustic analysis — 1. severity and character of dysphonia (measured by Auditory Perceptual Assessment using a modified GRBAS scale which gives scores as regard the degree and severity of dysphonia and its character.
  2. Acoustic Analysis of voice : which is Computerized Speech Laboratory analysis of voice that gives the following measures jitter (%), shimmer (dB), and harmonic to noise ratio (H/N).
  3. the degree of social ,emotional ,functional and physical disturbance ,if present in those children with voice disorders by application of The Arabic Pediatric Voice Related Quality of Life (PV-RQOL).

SUMMARY:
The aim of this study is to assess the Correlation between The Arabic Pediatric Voice Related Quality of Life (PV-RQOL), The Auditory Perceptual Assessment and Acoustic Analysis of voice of dysphonic children. This is important to provide an efficient therapeutic strategy for these children.

DETAILED DESCRIPTION:
Voice is the carrier wave for speech signal. It can also be defined as an audible sound produced by phonation . It is a primary mean of expression and oral communication and has life-long importance to social well-being.

Through life, voice development follows and represents organic, psychological, and social changes in the person .

Any disruption of the function of voice is called dysphonia . defination of dysphonia is perceptual audible change of a patient's habitual voice as self-judged or judged by his or her listeners.

The incidence of the pediatric voice disorders ranges from 6%-23%, while, stated that voice disorders affect approximately 6-9% of pediatric population. Boys were statistically more likely to have dysphonia (7.5%) over girls (4.6%) , abnormal vocal presentations (symptomatology) include: phonasthenia ,dysphonia, aphonia and dysodia. Dysphonia may adversely impact a child's general health, communicative effectiveness, social and educational development, self-esteem, and participation in school group activities. Hence, dysphonia has a substantial negative effect on children's lives.Although voice disorders are common in the pediatric population; there is still a lack of information available to clinicians regarding evaluation and treatment of pediatric voice disorders.

Etiology of Voice disorders can be subdivided into 3 main groups: There are the organic voice disorders (There are detectable morphological changes in the vocal apparatus), Non-organic (functional) voice disorders (There is no detectable organic pathology in the structure of the larynx) and Minimal Associated Pathological Lesions (MAPLs) (Long-standing, non-organic (functional) voice disorders leading to the creation of detectable organic changes.

The protocol of evaluation of voice disorders is constructed /built in escalating stepwise stages from the simple subjective bed-side diagnostic procedures to the more sophisticated objective quantitative instrumental measures. Thus the protocol encompasses the following 3 levels which are 1- Elementary diagnostic procedures, 2-Clinical diagnostic aids 3-Additional instrumental measures .

Several instruments have been designed specifically to evaluate quality of life outcomes in dysphonic populations. The best validated and most utilized surveys are the Voice Handicap Index (VHI) , the Voice Outcome Survey (VOS) and the Voice-Related Quality of Life (V-RQoL) . These instruments were designed to be used in the assessment of dysphonic patients and were validated in adult populations. Since their dissemination, each of these instruments have produced a pediatric analogue, namely a pediatric VOS (PVOS) , a pediatric V-RQoL and a pediatric VHI (PVHI).

Questionnaire may help to increase the patient's awareness of the impact of dysphonia and his motivation for change. The Questionnaires have also been proven sensitive to post-changes and are an additional and valuable tool in the determination of therapy efficiency.

At Minia University, a study was carried out to develop an Arabic version of PVRQoL and test its validity and reliability .The results suggested that the APVRQoL is a valid and reliable assessment tool that can be used by the parents of Arabic-speaking children or by the children themselves (when they are older) with voice disorders to assess the impact of dysphonia on the quality of their lives.

The (PV-RQOL) has 10 questions that are divided among 4 subdomains: The social (questions no: 8 and 10), emotional (questions no: 4 and 5) , The physical (questions no: 2 and 3) and the functional (questions no: 1, 6,7 and 9), each question is rated from 1to5 (1=no problem and is given"10 points",2=a small amount and is given"7.5points",3=a moderate amount and is given"5 points",4=a lot and is given"2.5 points", and 5=problem is as bad as it can be, and is given"0 points". Thus the raw scores can range from 0 to 100 points with higher scores indicating a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

-clinical diagnosis of change of voice due to functional (non-organic) causes or due to Minimal Associated Pathological Lesions (MAPLs).

Exclusion Criteria:

* Mental Retardation.
* chronic illnesses affecting their quality of lives.
* organic voice disorders.

Ages: 6 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: One hundred twenty six (126) children will participate in the study; in 2 groups ,1-study group 63 children they have dysphonia due to functional (non-organic) causes or due to Minimal Associated Pathological Lesions (MAPLs),2-control group 63 children without vocal complaints They will be recruited from the outpatient clinic of Phoniatric Unit, Assiut University Hospital.
  Participants (whether their caretakers or themselves) will sign an informed consent of approval to participate in the study after explanation of the study procedures.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
All participants' scores of (PV-RQOL) questionnaire will be correlated with scores of auditory perceptual assessment and Acoustic voice analysis. | baseline
  Application of the Arabic Pediatric Voice Related Quality of Life (PV-RQOL): all participants /parents of the participants will be given (PV-RQOL) form that consists of 10 questions divided among 4 subdomains: The social (questions no: 8 and 10), emotional (questions no: 4 and 5) , The physical (questions no: 2 and 3) and the functional (questions no: 1, 6,7 and 9) . Thus the total score can range from 0 to 100 points with higher scores indicating a better quality of life.and Auditory perceptual assessment (APA) of the participant's voice: the domains will be graded on a scale of 0-3, in which 0 is normal and 3 is severe.and Acoustic voice analysis: will be carried out using Kay Elemetrics' Computerized Speech Laboratory. These measures will be obtained by recording the voice of each participant using a microphone positioned ∼10 cm from his/her mouth and the participantswill be asked to phonate a sustained vowel /a/ at comfortable pitch and intensity levels.

REFERENCES:
- [Background] Lopes LW, Barbosa Lima IL, Alves Almeida LN, Cavalcante DP, de Almeida AA. Severity of voice disorders in children: correlations between perceptual and acoustic data. J Voice. 2012 Nov;26(6):819.e7-12. doi: 10.1016/j.jvoice.2012.05.008. PMID 23177753
- [Background] Kotby MN, Shiromoto O, Hirano M. The accent method of voice therapy: effect of accentuations on FO, SPL, and airflow. J Voice. 1993 Dec;7(4):319-25. doi: 10.1016/s0892-1997(05)80120-1. PMID 8293064
- [Background] Carding PN, Roulstone S, Northstone K; ALSPAC Study Team. The prevalence of childhood dysphonia: a cross-sectional study. J Voice. 2006 Dec;20(4):623-30. doi: 10.1016/j.jvoice.2005.07.004. Epub 2005 Dec 19. PMID 16360302
- [Background] Trani M, Ghidini A, Bergamini G, Presutti L. Voice therapy in pediatric functional dysphonia: a prospective study. Int J Pediatr Otorhinolaryngol. 2007 Mar;71(3):379-84. doi: 10.1016/j.ijporl.2006.11.002. Epub 2006 Nov 29. PMID 17137639
- [Background] Blumin JH, Keppel KL, Braun NM, Kerschner JE, Merati AL. The impact of gender and age on voice related quality of life in children: normative data. Int J Pediatr Otorhinolaryngol. 2008 Feb;72(2):229-34. doi: 10.1016/j.ijporl.2007.10.015. Epub 2007 Dec 11. PMID 18063123
- [Background] Connor NP, Cohen SB, Theis SM, Thibeault SL, Heatley DG, Bless DM. Attitudes of children with dysphonia. J Voice. 2008 Mar;22(2):197-209. doi: 10.1016/j.jvoice.2006.09.005. Epub 2007 May 18. PMID 17512168
- [Background] Gliklich RE, Glovsky RM, Montgomery WW. Validation of a voice outcome survey for unilateral vocal cord paralysis. Otolaryngol Head Neck Surg. 1999 Feb;120(2):153-8. doi: 10.1016/S0194-5998(99)70399-2. PMID 9949345
- [Background] Hartnick CJ. Validation of a pediatric voice quality-of-life instrument: the pediatric voice outcome survey. Arch Otolaryngol Head Neck Surg. 2002 Aug;128(8):919-22. doi: 10.1001/archotol.128.8.919. PMID 12162771
- [Background] Boseley ME, Cunningham MJ, Volk MS, Hartnick CJ. Validation of the Pediatric Voice-Related Quality-of-Life survey. Arch Otolaryngol Head Neck Surg. 2006 Jul;132(7):717-20. doi: 10.1001/archotol.132.7.717. PMID 16847178
- [Background] Zur KB, Cotton S, Kelchner L, Baker S, Weinrich B, Lee L. Pediatric Voice Handicap Index (pVHI): a new tool for evaluating pediatric dysphonia. Int J Pediatr Otorhinolaryngol. 2007 Jan;71(1):77-82. doi: 10.1016/j.ijporl.2006.09.004. Epub 2006 Oct 13. PMID 17046072
- [Background] Verduyckt I, Remacle M, Jamart J, Benderitter C, Morsomme D. Voice-related complaints in the pediatric population. J Voice. 2011 May;25(3):373-80. doi: 10.1016/j.jvoice.2009.11.008. Epub 2010 Apr 1. PMID 20359863